CLINICAL TRIAL: NCT05172050
Title: Multicenter, Adaptive, Randomized, Placebo-controlled, Double Blind, Parallel-group Phase 2/3 Trial, to Study Efficacy and Safety of Two Doses of Raloxifene in Adult Paucisymptomatic COVID-19 Patients.
Brief Title: Multicenter Double Blind, Parallel-group Phase 2/3 Trial, to Study Raloxifene in Adult COVID-19 Patients.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dompé Farmaceutici S.p.A (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLX0120; 2020-003936-25 (EudraCT Number)
Record Dates: First submitted 2021-12-23; First posted 2021-12-29 (Actual); Results first posted 2023-12-14 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2022-06

CONDITIONS: SARS CoV 2 Infection
Keywords: COVID-19; SARS-CoV-2; severe pneumonia; pneumonia
MeSH Terms: conditions — COVID-19; Pneumonia | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Intervention Model Description: Multicenter, adaptive, double-blind, randomized, placebo controlled, double blind, parallelgroup, to study efficacy and safety, with the following adaptive components:
  * Parallel multi-arms (2 interventional arms and 1 placebo control arm);
  * A 2-stage sequential design (1 interim analysis + 1 final analysis);
  * Sample size re-calculation at interim stage;
  * Stopping rule for efficacy or futility at interim stage.
Who Masked: Participant, Investigator
Masking Description: Appearance, including packaging and labelling, of the investigational medicinal product (IMP, capsules, packaging) will not allow to recognize actual treatment (either raloxifene or placebo).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Raloxifene 60 mg (Experimental): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing 60 mg of the active substance or placebo), a single daily oral dose of raloxifene 60 mg was administered; the treatment was taken by the patients for two weeks.
  Interventions: Drug: Raloxifene
- Group 2: Raloxifene 120 mg (Experimental): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing 60 mg of the active substance or placebo), a single daily oral dose of raloxifene 120 mg was administered; the treatment was taken by the patients for two weeks.
  Interventions: Drug: Raloxifene
- Group 3: Placebo. (Placebo Comparator): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing placebo), a single daily oral dose of placebo (2 capsules guarantee the blinding design) was administered; the treatment was taken by the patients for two weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Raloxifene — Raloxifene was administered as 60 mg hard gelatine capsule(s) once a day. Starting from day 2 of treatment: one single capsule (plus one of placebo to guarantee the blinding) containing 60 mg raloxifene was administered in Group 1, and 2 capsules 60 mg each for a total of 120 mg in Group 2.
  Arms: Group 1: Raloxifene 60 mg; Group 2: Raloxifene 120 mg
Other: Placebo — Placebo was administered orally once a day as 2 capsules (for maintaining the blinding design)
  Other Names: control
  Arms: Group 3: Placebo.

SUMMARY:
The objective of the study is to evaluate the efficacy and safety of two different doses of raloxifene orally administered compared to placebo in patients with early diagnosis of paucisymptomatic COVID-19.

Primary objectives:

* Evaluation of the effectiveness of therapy in reducing the proportion of subjects who still have viruses in the upper airways after 7 days of therapy
* Evaluation of the effectiveness of therapy in reducing the proportion of subjects who requires supplemental oxygen therapy and/or mechanical ventilation within 14 days of starting therapy

Secondary objectives:

* Evaluation of the effectiveness of therapy in reducing the proportion of subjects who still have viruses in the upper airways after 14 and 28 days of therapy
* Evaluation of the effectiveness of therapy in reducing the proportion of subject patients who requires supplemental oxygen therapy and/or mechanical ventilation within 7 or 28 days of starting therapy
* 7, 14 and 28 days drug safety and tolerability profile
* Assessment of body temperature, blood and biochemical parameters between T0 and T28

DETAILED DESCRIPTION:
The study is a phase 2/3, multicenter, adaptive, randomized, placebo-controlled, double blind, parallel-group study to evaluate efficacy and safety of two doses of raloxifene in adult paucisymptomatic COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subject autonomously provides informed consent prior to initiation of any study procedures
2. Males and females ≥ 40 years old
3. Understands and agrees to comply with planned study procedures, has the availability of an email address as well as an Internet connection at domicile location
4. Agrees to the collection of nasopharyngeal swabs and venous blood samples per protocol
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by an approved molecular test (PCR) in Europe within 10 days at the screening time
6. Patient paucisymptomatic who complains at the screening time at least one of the following symptoms mild to moderate: fever, dyspnea, headache, cough, dysgeusia, conjunctivitis, vomiting, diarrhea, anosmia, muscle or body aches or other symptoms which in the opinion of the Investigator are part of the COVID-19 clinical picture
7. No need of supplemental oxygen therapy, mechanical ventilation
8. Females of child-bearing potential and with an active sexual life must not wish to get pregnant within 30 days after the end of the study and must be using at least one of the following reliable methods of contraception:

   1. Hormonal contraception, systemic, implantable, transdermal, or injectable contraceptives for at least 2 months before the screening visit until 30 days after final visit
   2. A non-hormonal intrauterine device [IUD] or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit until 30 days after final visit
   3. A male sexual partner who agrees to use a male condom with spermicide
   4. A sterile sexual partner

Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted. For all female subjects, with child-bearing potential, pregnancy test result must be negative before first drug intake on T7 and T14.

Exclusion Criteria:

1. Being totally asymptomatic at the screening time
2. Requires supplemental oxygen therapy or mechanical ventilation
3. Being already under raloxifene or other SERM treatment for another medical condition at the time of randomization
4. Being concurrently involved in another trial with IP or participation in any clinical trial with IP for 1 months before this study. The 1-month interval is calculated as the time between the last visit of the previous study and the first day of the present study (date of the informed consent signature)
5. Clinically significant abnormal physical findings which could interfere with the objectives of the study
6. Diseases:

   1. history of stroke and/or venous thromboembolism;
   2. known moderate / severe renal impairment: Chronic Kidney Disease (CKD) stage 3 or higher;
   3. known liver disease (Child-Pugh Class A or higher);
   4. presence of known hypoalbuminemia;
   5. endometrial bleeding;
   6. signs or symptoms of endometrial cancer
7. Autoimmune diseases receiving therapy at the time of randomization
8. Risk of venous thrombosis or any condition/disease that could bring to an extended period of immobilization
9. Ascertained or presumptive hypersensitivity to the active principles (raloxifene) and/or excipients or allergic reactions in general, which the Investigator considers may affect the outcome of the study
10. Medications: in particular cholestyramine (or any ion exchange resin), medications used in treatment of early or advanced breast cancer (including adjuvant therapy), warfarin, any drug that cannot be coadministered with the experimental compound
11. Pregnancy:

    1. positive or missing pregnancy test before first drug intake or day 1;
    2. pregnant or lactating women;
12. Women of childbearing potential and fertile men who does not agree to use at least one primary form of contraception for the duration of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-01-22 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sergio, MD, PhD, Study Director — Dompé Farmaceutici
Locations (11):
- France (4):
  - CHU Amiens, Amiens
  - Clinique de l'infirmerie protestante de Lyon, Caluire-et-Cuire
  - CH Emile Roux le Puy en Velay, Le Puy-en-Velay
  - Centre Hospitalier de Troyes, Troyes
- Italy (6):
  - Humanitas Gavazzeni, Bergamo
  - Ospedale San Salvatore, L’Aquila
  - AO dei Colli (Ospedale Monaldi), Napoli
  - INMI Lazzaro Spallanzani, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A.O.U. Città della Salute e della Scienza, Torino
- Hospital Universitario Virgen de la Victoria, Málaga, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicastri E, Marinangeli F, Pivetta E, Torri E, Reggiani F, Fiorentino G, Scorzolini L, Vettori S, Marsiglia C, Gavioli EM, Beccari AR, Terpolilli G, De Pizzol M, Goisis G, Mantelli F, Vaia F, Allegretti M; Raloxifene Territorial Health COVID19 STUDY GROUP. A phase 2 randomized, double-blinded, placebo-controlled, multicenter trial evaluating the efficacy and safety of raloxifene for patients with mild to moderate COVID-19. EClinicalMedicine. 2022 Jun;48:101450. doi: 10.1016/j.eclinm.2022.101450. Epub 2022 May 12. PMID 35582123

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Actual recruitment was greatly slower than expected and this determined a significant delay in study conduction, which in turn reflected on a study completion forecast that was not in line with Sponsor's planning.
Pre-assignment Details: Due to the premature study interruption, the sample size was smaller than that originally planned due to several reason that caused difficulties in patients enrolment.
Period: Overall Study
Arm/Group | Group 1: Raloxifene 60 mg | Group 2: Raloxifene 120 mg | Group 3: Placebo.
Started | 22 | 20 | 19
Full Analysis Set Population (FAS) | 22 | 20 | 19
Per-Protocol Population (PP) | 18 | 17 | 17
Safety Population (SAF) | 22 | 20 | 19
Completed (treatment completion) | 10 | 9 | 8
Not Completed | 12 | 11 | 11
Not completed — Negative Nasopharyngeal swab | 5 | 5 | 3
Not completed — Development of AE or unacceptable toxicity | 5 | 4 | 7
Not completed — Other | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) population included all randomized patients who received at least one dose of the study medication. The FAS population was used for demographics, and primary and secondary efficacy analyses
Groups:
- Raloxifene 60 mg (FAS): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing 60 mg of the active substance or placebo), a single daily oral dose of raloxifene 60 mg was administered; the treatment was taken by the patients for two weeks.
  Raloxifene: Raloxifene was administered as 60 mg hard gelatine capsule(s) once a day. Starting from day 2 of treatment: one single capsule (plus one of placebo to guarantee the blinding) containing 60 mg raloxifene was administered in Group 1, and 2 capsules 60 mg each for a total of 120 mg in Group 2.
- Raloxifene 120 mg (FAS): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing 60 mg of the active substance or placebo), a single daily oral dose of raloxifene 120 mg was administered; the treatment was taken by the patients for two weeks.
  Raloxifene: Raloxifene was administered as 60 mg hard gelatine capsule(s) once a day. Starting from day 2 of treatment: one single capsule (plus one of placebo to guarantee the blinding) containing 60 mg raloxifene was administered in Group 1, and 2 capsules 60 mg each for a total of 120 mg in Group 2.
- Placebo (FAS): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing placebo), a single daily oral dose of placebo (2 capsules guarantee the blinding design) was administered; the treatment was taken by the patients for two weeks.
  Placebo: Placebo was administered orally once a day as 2 capsules (for maintaining the blinding design)
- Total: Total of all reporting groups
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS) | Total
Number analyzed (Participants) | 22 | 20 | 19 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 15 | 15 | 48
  >=65 years | 4 | 5 | 4 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.88) | 58.9 (10.03) | 54.6 (9.33) | 56.2 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 9 | 28
  Male | 11 | 12 | 10 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 22 | 20 | 19 | 61
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 22 | 20 | 19 | 61

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Undetectable SARS-CoV-2 at PCR at Day 7 After Randomization in the FAS
Description: Number of participants who, after an approved molecular test (PCR), were not detected as SARS-CoV2 positive. Based on Approved molecular test (PCR) result at day 7, the responses were considered as "detectable" if PCR result was "Positive" otherwise "undetectable" if PCR result was "Negative" .
Time Frame: At Day 7
Population: The Full Analysis Set (FAS) population included all randomized patients who received at least one dose of the study medication. The FAS population was used for primary and secondary efficacy analyses.
Measure: Count of Participants; unit: Participants
Groups:
- Raloxifene 60 mg: After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing 60 mg of the active substance or placebo), a single daily oral dose of raloxifene 60 mg was administered; the treatment was taken by the patients for two weeks.
  Raloxifene: Raloxifene was administered as 60 mg hard gelatine capsule(s) once a day. Starting from day 2 of treatment: one single capsule (plus one of placebo to guarantee the blinding) containing 60 mg raloxifene was administered in Group 1, and 2 capsules 60 mg each for a total of 120 mg in Group 2.
- Raloxifene 120 mg: After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing 60 mg of the active substance or placebo), a single daily oral dose of raloxifene 120 mg was administered; the treatment was taken by the patients for two weeks.
  Raloxifene: Raloxifene was administered as 60 mg hard gelatine capsule(s) once a day. Starting from day 2 of treatment: one single capsule (plus one of placebo to guarantee the blinding) containing 60 mg raloxifene was administered in Group 1, and 2 capsules 60 mg each for a total of 120 mg in Group 2.
- Placebo: After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing placebo), a single daily oral dose of placebo (2 capsules guarantee the blinding design) was administered; the treatment was taken by the patients for two weeks.
  Placebo: Placebo was administered orally once a day as 2 capsules (for maintaining the blinding design)
Arm/Group | Raloxifene 60 mg | Raloxifene 120 mg | Placebo
Number analyzed (Participants) | 22 | 20 | 19
Participants | 7 | 4 | 0
Statistical Analysis 1: Comparison: Raloxifene 60 mg vs Placebo; Test type: Superiority — Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; p = 0.0109, Regression, Logistic; Odds Ratio (OR) = 9.990, 95% CI 2-sided [lower limit 1.781] (Upper limit is not estimable (NE) due to the low number of events)
Statistical Analysis 2: Comparison: Raloxifene 120 mg vs Placebo; Test type: Superiority — Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; p = 0.0673, Regression, Logistic; Odds Ratio (OR) = 5.414, 95% CI 2-sided [lower limit 0.858] (The upper limit is not estimable (NE), due to the low number of events)
Statistical Analysis 3: Comparison: Raloxifene 60 mg vs Placebo; This sensitivity analysis is conducted on the per protocol (PP) population: n=18 in the Raloxifene 60 mg arm; n=17 in the Raloxifene 120 mg arm; and n=17 in the Placebo arm; Test type: Superiority; p = 0.0061, Regression, Logistic — Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 12.186, 95% CI 2-sided [lower limit 2.147] (The upper limit was not estimable due to the low number of events)
Statistical Analysis 4: Comparison: Raloxifene 120 mg vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0567, Regression, Logistic — Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 5.936, 95% CI 2-sided [lower limit 0.938] (The upper limit was not estimable due to the low number of events)

2. Primary Outcome: Number of Participants Not Requiring Oxygen Therapy and/or Mechanical Ventilation at Day 14 After Randomization in the FAS
Description: Proportion of participants who does not require supplemental oxygen therapy (NEWS ≤ 2) and/or mechanical ventilation. NEWS is a system for scoring the physiological measurements that are routinely recorded at the patient's bedside. NEWS uses six physiological measurements. An additional two points are added if the patient is receiving oxygen therapy. The total possible score ranges from 0 to 20. If collected NEWS score > 2 or mechanical ventilation with result "Yes" then the response was considered as "Required". If collected NEWS score ≤ 2 and mechanical ventilation with result "No" then the response was considered as "Not Required" (if both NEWS score and mechanical ventilation were missing, patient was considered as missing).
Time Frame: At Day 14
Population: The Full Analysis Set (FAS) population included all randomized patients who received at least one dose of the study medication. The FAS population was used for primary and secondary efficacy analyses;
Measure: Count of Participants; unit: Participants
Arm/Group | Raloxifene 60 mg | Raloxifene 120 mg | Placebo
Number analyzed (Participants) | 22 | 20 | 19
Participants | 10 | 8 | 8
Statistical Analysis 1: Comparison: Raloxifene 60 mg vs Placebo; Test type: Superiority — Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; p = 0.7121, Regression, Logistic; Odds Ratio (OR) = 1.663, 95% CI 2-sided [0.337 to 9.053]
Statistical Analysis 2: Comparison: Raloxifene 120 mg vs Placebo; Test type: Superiority — Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; p > 0.999, Regression, Logistic; Odds Ratio (OR) = 0.963, 95% CI 2-sided [0.185 to 4.977]
Statistical Analysis 3: Comparison: Raloxifene 60 mg vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.5378, Regression, Logistic — Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 2.340, 95% CI 2-sided [0.350 to 20.153]
Statistical Analysis 4: Comparison: Raloxifene 120 mg vs Placebo; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p > 0.999, Regression, Logistic — Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 1.209, 95% CI 2-sided [0.185 to 8.589]

3. Secondary Outcome: Number of Participants With Undetectable SARS-CoV-2 at PCR at Days 14 and 28 After Randomization in the FAS
Description: Number of participants with undetectable SARS-CoV-2 at PCR at day 14 after randomization, and at day 28 after randomization. Based on Approved molecular test (PCR) result at days 14 and 28 after randomization, the responses were considered as "detectable" if PCR result was "Positive" otherwise "undetectable" if PCR result was "Negative".
Time Frame: At days 14 and 28 after randomization
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
Participants
  at Day 14 | 10 | 14 | 7
  at Day 28 | 17 | 17 | 12
Statistical Analysis 1: Comparison: Raloxifene 60 mg (FAS) vs Placebo (FAS); at Day 14; Test type: Superiority; p > 0.999, Regression, Logistic; Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 1.114, 95% CI 2-sided [0.219 to 5.708]
Statistical Analysis 2: Comparison: Raloxifene 120 mg (FAS) vs Placebo (FAS); At day 14; Test type: Superiority; p = 0.2553, Regression, Logistic; Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 3.202, 95% CI 2-sided [0.541 to 22.116]
Statistical Analysis 3: Comparison: Raloxifene 60 mg (FAS) vs Placebo (FAS); at Day 28; Test type: Superiority; p = 0.6189, Regression, Logistic; Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 2.160, 95% CI 2-sided [0.294 to 18.532]
Statistical Analysis 4: Comparison: Raloxifene 120 mg (FAS) vs Placebo (FAS); at Day 28; Test type: Superiority; p = 0.1662, Regression, Logistic; Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 7.220, 95% CI 2-sided [0.586 to 413.499]

4. Secondary Outcome: Number of Participants Not Requiring Oxygen Therapy and/or Mechanical Ventilation at Day 7 an d at Day 28 in the FAS
Description: Proportion of participants who does not require supplemental oxygen therapy (NEWS ≤ 2) and/or mechanical ventilation after randomization;
Time Frame: At days 7 and 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
Participants
  at Day 7 | 12 | 12 | 11
  at Day 28 | 9 | 12 | 7
Statistical Analysis 1: Comparison: Raloxifene 60 mg (FAS) vs Placebo (FAS); at Day 7; Test type: Superiority; p > 0.999, Regression, Logistic; Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 0.972, 95% CI 2-sided [0.193 to 4.906]
Statistical Analysis 2: Comparison: Raloxifene 120 mg (FAS) vs Placebo (FAS); at Day 7; Test type: Superiority; p > 0.999, Regression, Logistic; Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 1.156, 95% CI 2-sided [0.200 to 6.822]
Statistical Analysis 3: Comparison: Raloxifene 60 mg (FAS) vs Placebo (FAS); at Day 28; Test type: Superiority; p > 0.999, Regression, Logistic; Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 1.066, 95% CI 2-sided [0.208 to 5.478]
Statistical Analysis 4: Comparison: Raloxifene 120 mg (FAS) vs Placebo (FAS); at Day 28; Test type: Superiority; p = 0.5465, Regression, Logistic; Analysis is based on Exact Binary logistic regression model with treatment group, age group and status as main effects; Odds Ratio (OR) = 2.068, 95% CI 2-sided [0.369 to 12.580]

5. Secondary Outcome: Number of Patients in Each National Early Warning Score (NEWS) Category in the FAS
Description: Proportion of patients in each National Early Warning Score (NEWS) category after randomization. NEWS is a system for scoring the physiological measurements that are routinely recorded at the patient's bedside. NEWS uses six physiological measurements: respiratory rate; oxygen saturation; temperature; systolic blood pressure; heart rate and level of consciousness. Each scores 0-3 and individual scores are added together for an overall score. An additional two points are added if the patient is receiving oxygen therapy. The total possible score ranges from 0 to 20. The higher the score, the worse the outcome.
Time Frame: At days 7, 14, 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
Participants
  Day 7 - Score 0 | 6 | 5 | 6
  Day 7 - Score 1 | 3 | 4 | 5
  Day 7 - Score 2 | 3 | 3 | 0
  Day 7 - Score 3 | 1 | 2 | 0
  Day 7 - Score 4 | 2 | 0 | 3
  Day 7 - Score 5 | 1 | 1 | 0
  Day 7 - Score 7 | 2 | 1 | 0
  Day 7 - Missing | 4 | 4 | 5
  Day 14 - Score 0 | 5 | 4 | 5
  Day 14 - Score 1 | 5 | 2 | 3
  Day 14 - Score 2 | 1 | 3 | 0
  Day 14 - Score 3 | 1 | 5 | 2
  Day 14 - Score 4 | 2 | 1 | 1
  Day 14 - Score 5 | 0 | 0 | 1
  Day 14 - Score 6 | 1 | 0 | 1
  Day 14 - Missing | 7 | 5 | 6
  Day 28 - Score 0 | 5 | 8 | 5
  Day 28 - Score 1 | 4 | 5 | 3
  Day 28 - Score 2 | 1 | 0 | 1
  Day 28 - Score 3 | 0 | 0 | 1
  Day 28 - Score 4 | 2 | 0 | 1
  Day 28 - Missing | 10 | 7 | 8

6. Secondary Outcome: Mean Value of National Early Warning Score (NEWS) Category in the FAS
Description: Mean value of National Early Warning Score (NEWS) category after randomization. NEWS is a system for scoring the physiological measurements that are routinely recorded at the patient's bedside. The total possible score ranges from 0 to 20. The higher the score the greater the clinical risk. Higher scores indicate the need for escalation, medical review and possible clinical intervention and more intensive monitoring
Time Frame: At days 7, 14, 28 after randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
score on a scale
  Day 7: number analyzed (Participants) | 18 | 16 | 14
  Day 7 | 2.2 (2.36) | 1.8 (1.98) | 1.2 (1.58)
  Day 14: number analyzed (Participants) | 15 | 15 | 13
  Day 14 | 1.6 (1.84) | 1.8 (1.37) | 1.8 (2.12)
  Day 28: number analyzed (Participants) | 12 | 13 | 11
  Day 28 | 1.2 (1.47) | 0.4 (0.51) | 1.1 (1.38)

7. Secondary Outcome: Number of Hospitalized Participants Who at the Beginning of the Study Were at Domicile Isolation After Randomization in the FAS
Description: Proportion of hospitalized participants at Day 7, Day 14 and Day 28 after randomization among subjects who at the beginning of the study were at domicile isolation.
Time Frame: At days 7, 14, 28
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
Participants
  Day 7 | 20 | 18 | 15
  Day 14 | 20 | 18 | 15
  Day 28 | 20 | 18 | 16
Statistical Analysis 1: Comparison: Raloxifene 60 mg (FAS) vs Placebo (FAS); The proportion of hospitalized participants who at the beginning of the study were at domicile isolation at Day 7, Day 14 and Day 28 after randomization was analysed using comparison of proportions (i.e. comparisons of each active treatment group versus placebo at each assessment day) through Fisher's exact test and was summarized using frequency and percent by treatment and visit. Herein Day 7 R60 vs Placebo; Test type: Superiority; p = 0.3899, Fisher Exact — P-Value comparing % among treatment groups Raloxifene 60mg versus Placebo using Fisher's Exact test
Statistical Analysis 2: Comparison: Raloxifene 120 mg (FAS) vs Placebo (FAS); The proportion of hospitalized participants who at the beginning of the study were at domicile isolation at Day 7, Day 14 and Day 28 after randomization was analysed using comparison of proportions (i.e. comparisons of each active treatment group versus placebo at each assessment day) through Fisher's exact test and was summarized using frequency and percent by treatment and visit. Herein Day 7 R120 vs placebo; Test type: Superiority; p = 0.4075, Fisher Exact — P-Value comparing % among treatment groups Raloxifene 120 mg versus Placebo using Fisher's Exact test
Statistical Analysis 3: Comparison: Raloxifene 60 mg (FAS) vs Placebo (FAS); The proportion of hospitalized participants who at the beginning of the study were at domicile isolation at Day 7, Day 14 and Day 28 after randomization was analysed using comparison of proportions (i.e. comparisons of each active treatment group versus placebo at each assessment day) through Fisher's exact test and was summarized using frequency and percent by treatment and visit. Herein Day 14 R60 vs placebo; Test type: Superiority; p = 0.3899, Fisher Exact — P-Value comparing % among treatment groups Raloxifene 60mg versus Placebo using Fisher's Exact test
Statistical Analysis 4: Comparison: Raloxifene 120 mg (FAS) vs Placebo (FAS); The proportion of hospitalized participants who at the beginning of the study were at domicile isolation at Day 7, Day 14 and Day 28 after randomization was analysed using comparison of proportions (i.e. comparisons of each active treatment group versus placebo at each assessment day) through Fisher's exact test and was summarized using frequency and percent by treatment and visit. Herein Day 14 R120 vs placebo; Test type: Superiority; p = 0.4075, Fisher Exact; P-Value comparing % among treatment groups Raloxifene 120mg versus Placebo using Fisher's Exact test
Statistical Analysis 5: Comparison: Raloxifene 60 mg (FAS) vs Placebo (FAS); The proportion of hospitalized participants who at the beginning of the study were at domicile isolation at Day 7, Day 14 and Day 28 after randomization was analysed using comparison of proportions (i.e. comparisons of each active treatment group versus placebo at each assessment day) through Fisher's exact test and was summarized using frequency and percent by treatment and visit. Herein Day 28 R60 vs placebo; Test type: Superiority; p = 0.6846, Fisher Exact — P-Value comparing % among treatment groups Raloxifene 60mg versus Placebo using Fisher's Exact test
Statistical Analysis 6: Comparison: Raloxifene 120 mg (FAS) vs Placebo (FAS); The proportion of hospitalized participants who at the beginning of the study were at domicile isolation at Day 7, Day 14 and Day 28 after randomization was analysed using comparison of proportions (i.e. comparisons of each active treatment group versus placebo at each assessment day) through Fisher's exact test and was summarized using frequency and percent by treatment and visit. Herein Day 28 R120 vs placebo; Test type: Superiority; p = 0.6614, Fisher Exact — P-Value comparing % among treatment groups Raloxifene 120mg versus Placebo using Fisher's Exact test

8. Secondary Outcome: Number of Participants Admitted to Intensive Care After Randomization in the FAS
Description: Proportion of participants admitted to intensive care. Intensive care is a special medical treatment in which a patient who is dangerously ill is kept under constant observation, typically in a dedicated department of a hospital.
Time Frame: At days 7,14 ,28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
Participants
  Day 7 | 0 | 0 | 0
  Day 14 | 0 | 0 | 0
  Day 28 | 0 | 0 | 0

9. Secondary Outcome: Number of Survivors in the FAS
Description: Proportion of survivors after randomization. There were no events (i.e. deaths) in any treatment groups and thus the median overall survival could not be estimated. Overall survival was analysed according to the Kaplan-Meier method. Time to event curves were compared (i.e. comparisons of each active treatment group versus placebo) using log-rank test and estimates of hazard ratio were obtained using Cox proportional hazards model.
Time Frame: At days 7, 14, 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
Participants | 22 | 20 | 19
Statistical Analysis 1: Comparison: Raloxifene 60 mg (FAS) vs Placebo (FAS); Test type: Superiority; Log Rank; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [1.00 to 1.00]
Statistical Analysis 2: Comparison: Raloxifene 120 mg (FAS) vs Placebo (FAS); Test type: Superiority; Log Rank — p value= not estimable; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [1.00 to 1.00]

10. Secondary Outcome: Quality of Life Questionnaire (EQ-5D-5L) at 3 Months After Randomization - EQ-5D Descriptive System
Description: The EQ-5D-5L consists of: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The EQ-5D-5L system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the 5 dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the 5 dimensions can be combined into a 5-digit number describing the patient's health state. In the EQ VAS - quantitative measure of health outcome - the patient records a self-rates health on a vertical visual analogue scale (numbered from 0 to 100) which goes from 'Best imaginable health state' (100) to 'Worst imaginable health state' (0).
Time Frame: At month 3 After Randomization
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
Participants
  mobility -no problems in walking about | 18 | 12 | 15
  mobility - slight problems in walking about | 1 | 5 | 2
  mobility - moderate problems in walking about | 0 | 0 | 1
  mobility-severe problems in walking about | 0 | 0 | 0
  mobility - unable to walk about | 0 | 0 | 0
  self care - no problems washing or dressing myself | 18 | 17 | 18
  self care - slight problems washing or dressing myself | 0 | 0 | 0
  self care - moderate problems washing or dressing myself | 1 | 0 | 0
  self care - severe problems washing or dressing myself | 0 | 0 | 0
  self care - unable to wash or dress myself | 0 | 0 | 0
  usual activities - no problems doing my usual activities | 14 | 14 | 12
  usual activities - slight problems doing my usual activities | 3 | 3 | 5
  usual activities - moderate problems doing my usual activities | 1 | 0 | 1
  usual activities - severe problems doing my usual activities | 1 | 0 | 0
  usual activities - unable to do my usual activities | 0 | 0 | 0
  Pain/discomfort - no pain or discomfort | 17 | 13 | 15
  Pain/discomfort - slight pain or discomfort | 0 | 4 | 2
  Pain/discomfort - moderate pain or discomfort | 1 | 0 | 0
  Pain/discomfort - severe pain or discomfort | 1 | 0 | 1
  Pain/discomfort - extreme pain or discomfort | 0 | 0 | 0
  Anxiety / Depression - I am not anxious or depressed | 13 | 10 | 13
  Anxiety / Depression - I am slightly anxious or depressed | 1 | 5 | 4
  Anxiety / Depression - I am moderately anxious or depressed | 5 | 2 | 1
  Anxiety / Depression - I am severely anxious or depressed | 0 | 0 | 0
  Anxiety / Depression - I am extremely anxious or depressed | 0 | 0 | 0

11. Secondary Outcome: Quality of Life Questionnaire (EQ-5D-5L) at 3 Months After Randomization - EQ VAS
Description: as for outcome 10
Time Frame: At month 3 After Randomization
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Raloxifene 60 mg (FAS) | Raloxifene 120 mg (FAS) | Placebo (FAS)
Number analyzed (Participants) | 22 | 20 | 19
score on a scale | 85.6 (13.7) | 75.2 (21.9) | 84.1 (11.5)

ADVERSE EVENTS:
Time Frame: The specific period of time over wich adverse events data were collected was within Day 7, 14 and 28 after randomization
Description: An Adverse Event (AE) was defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which did not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to the medicinal product.
Groups:
- Raloxifene 60 mg (SAF): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing 60 mg of the active substance or placebo), a single daily oral dose of raloxifene 60 mg was administered; the treatment was taken by the patients for two weeks.
  Raloxifene: Raloxifene was administered as 60 mg hard gelatine capsule(s) once a day. Starting from day 2 of treatment: one single capsule (plus one of placebo to guarantee the blinding) containing 60 mg raloxifene was administered in Group 1, and 2 capsules 60 mg each for a total of 120 mg in Group 2.
- Raloxifene 120 mg (SAF): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing 60 mg of the active substance or placebo), a single daily oral dose of raloxifene 120 mg was administered; the treatment was taken by the patients for two weeks.
  Raloxifene: Raloxifene was administered as 60 mg hard gelatine capsule(s) once a day. Starting from day 2 of treatment: one single capsule (plus one of placebo to guarantee the blinding) containing 60 mg raloxifene was administered in Group 1, and 2 capsules 60 mg each for a total of 120 mg in Group 2.
- Placebo (SAF): After an administration of two oral doses in the first day of treatment (one dose in the morning and one dose in the evening, each dose administered with 2 capsules containing placebo), a single daily oral dose of placebo (2 capsules guarantee the blinding design) was administered; the treatment was taken by the patients for two weeks.
  Placebo: Placebo was administered orally once a day as 2 capsules (for maintaining the blinding design)
Arm/Group | Raloxifene 60 mg (SAF) | Raloxifene 120 mg (SAF) | Placebo (SAF)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20 | 0/19
Serious Adverse Events (participants affected / at risk) | 3/22 | 2/20 | 5/19
Other Adverse Events (participants affected / at risk) | 6/22 | 8/20 | 6/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raloxifene 60 mg (SAF) (N=22) | Raloxifene 120 mg (SAF) (N=20) | Placebo (SAF) (N=19)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raloxifene 60 mg (SAF) (N=22) | Raloxifene 120 mg (SAF) (N=20) | Placebo (SAF) (N=19)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 2 (2) | 1 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Lipids increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Pareaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Postmenopausal haemorrage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT05172050/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT05172050/SAP_001.pdf